CLINICAL TRIAL: NCT00891670
Title: Validation of Adjunctive Cilostazol According to CYP2C19 Polymorphism: Prospective, Randomized, Single-Center Trial:
Brief Title: Comparison of Platelet Inhibition With Adjunctive Cilostazol Versus High Maintenance-Dose Clopidogrel According to Hepatic Cytochrome 2C19 Allele (CYP2C19) Polymorphism
Acronym: ACCEL2C19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Young-Hoon Jeong, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCS-0901-D
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Stenosis; Maximal Platelet Aggregation; Late Platelet Aggregation; High Post-Treatment Platelet Reactivity
Keywords: CYP2C19 polymorphism; platelet; Adjunctive cilostazol; high maintenance dose clopidogrel; P2Y12 Reaction Unit
MeSH Terms: conditions — Coronary Stenosis | interventions — Cilostazol; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple group (Active Comparator): received cilostazol 100 mg twice daily in addition to aspirin 100mg and clopidogrel 75mg once daily
  Interventions: Drug: cilostazol; Drug: aspirin
- high maintenance dose group (Active Comparator): received clopidogrel 150 mg/day with aspirin 100mg once daily
  Interventions: Drug: clopidogrel; Drug: aspirin

INTERVENTIONS:
Drug: cilostazol — 100mg twice daily for at least 1 month
  Other Names: pletaal
  Arms: triple group
Drug: clopidogrel — 75mg once daily (triple group arm)
  150mg once daily (high maintenance dose group arm)
  Other Names: plavix
  Arms: high maintenance dose group
Drug: aspirin — aspirin 100mg

SUMMARY:
The purpose of this study was to determine the impact of adjunctive cilostazol on platelet inhibition in carriers and non-carriers of the loss-of-function CYP2C19 allele.

DETAILED DESCRIPTION:
The additional platelet inhibition with clopidogrel, a thienopyridine inhibitor of the platelet P2Y12 adenosine diphosphate (ADP) receptor, has reduced the risk of ischemic events after coronary stent implantation. Because of inter-individual variability in platelet response to clopidogrel, a significant proportion of suboptimal platelet inhibition has been reported. In addition, persistent residual platelet reactivity measured with platelet function testing has shown the association with the cardiovascular outcomes after percutaneous coronary intervention(PCI).

Various clinical factors and genetic polymorphisms have been studied to predict the degree of antiplatelet response to clopidogrel. Interestingly, recent studies found that carriers of the loss-of-function hepatic cytochrome (CYP) 2C19 allele had significantly lower levels of the active metabolite of clopidogrel, diminished platelet inhibition, and a higher rate of major adverse cardiovascular events than did non-carriers, in the setting of PCI and acute coronary syndrome(ACS). These findings raise the need of solutions to overcome enhanced post-clopidogrel platelet reactivity by the influence of the loss-of-function CYP2C19 allele. Increasing the dose of clopidogrel and new potent P2Y12 antagonists(such as prasugrel) may be alternative antiplatelet regimens in patients with the loss-of-function CYP variant.

Cilostazol reversibly induces platelet inhibition via its blockade of phosphodiesterase (PDE) type 3 and is catalysed mainly by CYP3A. A recent study demonstrated that adjunctive cilostazol to dual antiplatelet therapy (triple antiplatelet therapy) intensified platelet inhibition as compared with a high maintenance-dose (MD) of 150 mg/day. Therefore, triple antiplatelet therapy could also be an alternative antiplatelet therapy to improve platelet inhibition and clinical outcomes in carriers of CYP2C19 mutant allele.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age
2. Significant coronary artery stenosis (> 70% by visual estimate)
3. Elective coronary stent implantation

Exclusion Criteria:

1. Acute myocardial infarction
2. Hemodynamic instability active bleeding and bleeding diatheses
3. Oral anticoagulation therapy with warfarin,use of peri-procedural glycoprotein IIb/IIIa inhibitors
4. Contraindication to antiplatelet therapy
5. Left ventricular ejection fraction < 30%
6. Leukocyte count < 3,000/mm3, platelet count < 100,000/mm3
7. AST or ALT ≥ 3 times upper normal
8. Serum creatinine level ≥ 2.5 mg/dL
9. stroke within 3 months
10. Noncardiac disease with a life expectancy < 1 year
11. Inability to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of maximal platelet aggregation | 30 days

SECONDARY OUTCOMES:
Rate of high post-clopidogrel platelet reactivity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD, phD, Principal Investigator — Gyeong-Sang Natinal University Hospital
Locations (1):
- Gyeong-Sang National University Hospital, Jinju, Gyeong-Nam, South Korea

REFERENCES:
- [Derived] Jeong YH, Abadilla KA, Tantry US, Park Y, Koh JS, Kwak CH, Hwang JY, Gurbel PA. Influence of CYP2C19*2 and *3 loss-of-function alleles on the pharmacodynamic effects of standard- and high-dose clopidogrel in East Asians undergoing percutaneous coronary intervention: the results of the ACCEL-DOUBLE-2N3 study. J Thromb Haemost. 2013 Jun;11(6):1194-7. doi: 10.1111/jth.12200. No abstract available. PMID 23517020
- [Derived] Jeong YH, Kim IS, Park Y, Kang MK, Koh JS, Hwang SJ, Kwak CH, Hwang JY. Carriage of cytochrome 2C19 polymorphism is associated with risk of high post-treatment platelet reactivity on high maintenance-dose clopidogrel of 150 mg/day: results of the ACCEL-DOUBLE (Accelerated Platelet Inhibition by a Double Dose of Clopidogrel According to Gene Polymorphism) study. JACC Cardiovasc Interv. 2010 Jul;3(7):731-41. doi: 10.1016/j.jcin.2010.05.007. PMID 20650435